CLINICAL TRIAL: NCT05894525
Title: Cohort Survey on Acute Phase Safety in Persons With Underlying Diseases Considered to Be at High Risk of Severe COVID-19 by Using Vaccination Information
Brief Title: Post-Marketing Safety Study in Japan in Participants With High Risk of Severe Exacerbation of Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) mRNA-1273 COVID-19 Vaccine
Status: Completed | Type: Observational
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: mRNA-1273-P916
Record Dates: First submitted 2023-06-05; First posted 2023-06-08 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: SARS-CoV-2
Keywords: mRNA-1273; mRNA-1273 vaccine; SARS-CoV-2; SARS-CoV-2 Vaccine; Coronavirus; Virus Diseases; Messenger RNA; COVID-19; COVID-19 Vaccine; Moderna
MeSH Terms: conditions — Coronavirus Infections; Virus Diseases; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort 1: Participants received 2 doses of mRNA-1273 vaccine approximately 4 weeks apart.

SUMMARY:
The goal of this study is to assess the adverse events in the acute phase observed after vaccination with the mRNA-1273 vaccine in persons with underlying diseases who are considered to have a high risk of severe exacerbation specified in COVID-19.

DETAILED DESCRIPTION:
Data collected from the JDMC Claims Database between August 2020 to November 2021.

ELIGIBILITY:
Inclusion Criteria:

* Participants registered to receive the mRNA-1273 vaccine in the Pep Up vaccination history Database
* Participants who have a history of vaccination with the mRNA-1273 vaccine in the Pep-Up vaccination history Database and have underlying diseases. Data period for confirmation of presence/absence of underlying disease is August 2020 to November 2021.

Exclusion Criteria:

* Underlying diseases that were determined undetectable by the pre-screening of JMDC
* Participants who did not consent to the questionnaire

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population was selected from participants who were registered to receive the mRNA-1273 vaccine in the Pep Up vaccination history Database and those who met the definition of underlying disease based on the claim data for 6 months from August 2020 to November 2021.
Sampling Method: Non-Probability Sample
Enrollment: 8844 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2023-05-26 (Actual); Study Completion 2023-05-26 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Solicited Acute Adverse Events | Up to 8 days post vaccination

CONTACTS AND LOCATIONS:
Locations (1):
- CMIC Co. Ltd.,, Tokyo, Japan